CLINICAL TRIAL: NCT05336149
Title: Demineralized Whole-tooth vs Demineralized Particulate Dentin Grafts in Alveolar Ridge Preservation. a Randomized Controlled Trial.
Brief Title: Demineralized Whole-tooth vs Demineralized Particulate Dentin Grafts in Alveolar Ridge Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed AbdelRaouf Hussein, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42022
Record Dates: First submitted 2022-04-04; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-tooth dentin graft (Experimental): The extracted tooth will be prepared as whole-tooth dentin graft and inserted in the extraction socket.
  Interventions: Procedure: Alveolar ridge preservation using whole-tooth dentin graft
- Particulate dentin graft (Active Comparator): The extracted tooth will be prepared as particulate dentin graft and inserted in the extraction socket.
  Interventions: Procedure: Alveolar ridge preservation using particulate dentin graft

INTERVENTIONS:
Procedure: Alveolar ridge preservation using whole-tooth dentin graft — Minimally-traumatic extraction of non-restorable teeth then grafting with whole-tooth dentin graft
  Arms: Whole-tooth dentin graft
Procedure: Alveolar ridge preservation using particulate dentin graft — Minimally-traumatic extraction of non-restorable teeth then grafting with particulate dentin graft
  Arms: Particulate dentin graft

SUMMARY:
The aim of this trial is to compare whole-tooth vs particulate dentin for their effects in alveolar ridge preservation.

DETAILED DESCRIPTION:
Extraction of the teeth is still one of the most commonly undertaken procedures in dental practices due to various reasons that render the teeth non-restorable. Following extraction, replacing the lost teeth with a prosthetic alternative that provides for both optimal esthetics and function can be challenging due to the inevitable events of socket healing that results in the reduction in alveolar bone height and width. To overcome these limitations and provide for adequate ridge volume, different bone preservation or augmentation techniques can be utilized with different clinical applications.

Alveolar ridge preservation is a procedure that attempts to reduce bone dimensional changes that naturally take place following tooth extraction. To overcome this problem, various approaches using various grafting materials and/or covering membranes have been proposed with varied success. The extracted tooth is no longer considered as clinical waste, it has been explored as an appropriate source for autogenous graft substitute. This idea emerged due to the shared embryonic origin of bone and teeth as well as the similarities in chemical structure as dentin is composed of 30-35% organic part and 65-70% inorganic part in comparison to alveolar bone, with inorganic and organic parts of 35% and 65% respectively. Both whole-tooth and particulate forms has been utilized for alveolar ridge preservation or augmentation but the superiority of one form over the other is not yet clear.

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable tooth indicated for extraction
* single-rooted teeth
* Patients at least 18 years or older
* Motivated patients, agree to sign informed consent and complete the follow-up period

Exclusion Criteria:

* Pregnant females
* active infection at extraction site
* Smokers
* systemic conditions affecting healing (e.g. diabetes, medications as bisphosphonates...)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Alveolar bone width change in mm | 6 months
  Alveolar bone linear width will be measured at baseline at final cone beam computed tomography (CBCT) scans. The change in bone width will be calculated as the subtraction of final width from baseline width and will be expressed in millimetres.

SECONDARY OUTCOMES:
Alveolar bone height change in mm | 6 months
  Alveolar bone linear height will be measured at baseline at final cone beam computed tomography (CBCT) scans. The change in bone height will be calculated as the subtraction of final height from baseline height and will be expressed in millimetres.
Histological assessment | 6 months
  Bone samples from at least one control and one intervention site will be taken during implant placement using a trephine bur. Samples will be examined for new bone formation (Yes/no) and inflammatory response (Yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided